CLINICAL TRIAL: NCT03025776
Title: One vs. Two Hand Use After Stroke: Role of Task Requirements
Acronym: FSIFall2016
Status: Completed | Type: Observational
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Maureen Whitford, Assistant Professor, Cleveland State University
Other Study IDs: IRB-FY2016-332
Record Dates: First submitted 2016-12-14; First posted 2017-01-20 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- stroke: individuals chronic (> 6 months) post-stroke
  Interventions: Behavioral: Reaching; Behavioral: Kinematic collection while reaching
- age matched health controls: age matched (double sample size anticipated) healthy controls
  Interventions: Behavioral: Reaching

INTERVENTIONS:
Behavioral: Reaching — sitting reaching under various task conditions (size, speed, location)
Behavioral: Kinematic collection while reaching — sitting reaching under various task conditions (size, speed, location), told how many & which hand to use, kinematic data collected
  Groups: stroke

SUMMARY:
To further develop interventions, the investigators need a better understanding of which task requirements (i.e. size or weight of object, location in workspace, etc.) drive a person after stroke to use 2 hands (as opposed to 1), and how the severity of their injury impacts this relationship and compare this to reaching in age-matched healthy controls subjects. A better understanding of this relationship will promote more informed development of rehabilitative interventions. This study proposes to explore in people after stroke and healthy controls: i.) how specific functional tasks requirements relate to 1 vs. 2 handed use, and ii.) how stroke severity impacts this arm use. We are proposing to study 15 individuals more than 6 months after stroke in the CSU Motor Behavior Lab for a two x 3 hour session of task-related reaching in sitting and 33 age matched (double sample size) healthy controls. The investigators will systematically vary task requirements (i.e. object size or weight, location in workspace, etc.), and record use of 1 versus 2 hands using videotaping as well as recording of quality of arm movement (kinematics) and muscle activity (EMG) in both arms.

ELIGIBILITY:
Inclusion Criteria:

subjects post-stroke

* passive flexibility (i.e. passive range of motion) in both arms such that the elbows can be straightened within 15 degrees of normal and shoulders be flexed (lifted up) at least 90 degrees and the hand needs to be able to open at least 75% of the way
* Actively (of each subject's own accord/ability) they must be able to, without assist in sitting and standing: straighten each elbow within 15 degrees of full range of motion, lift each arm up at at least 60 degrees from at the side, open each hand from a gross grasp volitionally.
* able to lift a glass jar using 1 or 2 hands in sitting and standing 10" above the table top.
* able to come to CSU for two x 3 hour visits with or without assistance of their caregiver/significant other
* No arm/hand injury within the last 3 months. * Individuals with common visual deficits post-stroke (1 side partial visual field cut aka homonymous hemianopsia) will be included.

Healthy controls:

-age matched (double sample size); no known injury to arms within last 3 months, able to carry out experimental task, no neurologic diagnoses/perceptual or sensory deficits affecting arm movement

Exclusion Criteria:

* Individuals who have any additional/other neurologic condition (i.e. Parkinsons Disease, multiple sclerosis, spinal cord injury)
* severe perceptual neglect (tested using clock drawing test ).
* Any individual who cannot answer phone screen questions competently and/or follow simple 2 step commands during the in-person screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults > 18 years old chronic post-stroke with upper extremity paresis yet able to complete a reach-to-grasp task independently with their paretic arm healthy controls > 18 years old (as per above)
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Hand Use (qualitative analysis of how many hands, which hand used) via video | within 1st day session only (assessed w/i 2-3 hour session only)
upper extremity kinematics (peak velocity, index of curvature, total movement time) | within 2nd day session only (assessed w/i 2-3 hour session only)
  measured on Day 2 session using electromagnetic sensors

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States